CLINICAL TRIAL: NCT06781541
Title: Physical Activity and Disability Prevention in Postmenopausal Women
Acronym: PADP-Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gdansk University of Physical Education and Sport (Other)
Collaborators: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AWFiS/2024_5_ZO; without grant number (Other: Gdansk University of Physical Education and Sport)
Record Dates: First submitted 2024-12-12; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Metabolic Syndrome; Fall Risk; Sarcopenia in Elderly; Osteopenia, Osteoporosis; Cardiovascular Diseases; Dementia; Quality of Life Outcomes; Cognitive Ability, General
Keywords: Physical activity; aerobic capacity; mobility; cognitive functions; quality of life; disability; postmenopausal women; Physical fitness
MeSH Terms: conditions — Metabolic Syndrome; Bone Diseases, Metabolic; Cardiovascular Diseases; Dementia; Motor Activity | interventions — Nordic Walking; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Nordic Walking (Experimental): Training is about 60 minutes each time, 3 times a week, each interval of 1 or 2 days, a total of 12 weeks. The primary focus is on utilizing a specialized pole for engaging in cross-country walking. This regimen entails approximately 10 minutes of warmup exercises, followed by around 40 minutes of brisk walking, and concluding with a period of relaxation stretching lasting between 5 to 8 minutes.
  Interventions: Behavioral: Nordic walking
- Daily life (Experimental): The individuals engaged in routine daily tasks, while being advised against incorporating any supplementary physical exertion.
  Interventions: Behavioral: Daily life
- Strength training (Experimental): Strength training was conducted in the gym with progressively increasing resistance from 65% to 75% of the maximum weight (one-repetition maximum (1-RM)). Participants performed 10-13 repetitions of the exercise in one serie. The training was carried out in station form and consisted of 10-13 exercises. There were rest intervals of 60-90 seconds between exercises. As intended, the training was comprehensive, i.e. it affected the muscles of the arms, legs, torso, abdomen and chest.
  Interventions: Behavioral: Strength training
- Bungy Pump Exercises (Experimental): The training lasts approximately 60 minutes each time, 3 times a week, for a period of 12 weeks. The main emphasis is placed on the use of a specialist Bungy Pump pole. Bungy Pump training allows participants to combine aerobic and strength training. Bungy Pump poles contain a built-in shock absorber (RSA) in the form of an elastic band. The additional resistance generated by the stretched band increases the overall intensity of the exercise and increases calorie consumption. The program classes will include approximately 10 minutes of warm-up exercises, followed by approximately 40 minutes of brisk walking, and at the end a period of relaxation stretching lasting from 5 to 8 minutes.
  Interventions: Behavioral: Bungy Pump Exercises
- Functional general conditioning training (Experimental): Functional general conditioning training was carried out at home with individually adjusted resistance depending on age and health. Participants typically performed 10-13 repetitions of a given exercise. 30-second rest intervals were used between exercises. As intended, the training was comprehensive, i.e. including muscles of the arms, legs, trunk, abdomen, chest, balance and flexibility exercises. Basic training equipment was used during the training.
  Interventions: Behavioral: Functional general conditioning training

INTERVENTIONS:
Behavioral: Nordic walking — NW training sessions are conducted by a certified NW instructor leading participants in the outdoor forest of Gdansk. Training is about 60 minutes each time, 3 times a week, each interval of 1 or 2 days, a total of 12 weeks. Participants used professional Nordic Pole.
  Arms: Nordic Walking
Behavioral: Strength training — Strength training was conducted in the gym with progressively increasing resistance from 65% to 75% of the maximum weight (one-repetition maximum (1-RM)). Participants performed 10-13 repetitions of the exercise in one serie. The training was carried out in station form and consisted of 10-13 exercises. There were rest intervals of 60-90 seconds between exercises. As intended, the training was comprehensive, i.e. it affected the muscles of the arms, legs, torso, abdomen and chest.
  Arms: Strength training
Behavioral: Bungy Pump Exercises — Buny Pump training sessions are conducted by a certified BP instructor leading participants in the outdoor forest of Gdansk. Training is about 60 minutes each time, 3 times a week, a total of 12 weeks. Participants used professional Bungy Pump Pole.
  Arms: Bungy Pump Exercises
Behavioral: Daily life — The individuals engaged in routine daily tasks, while being advised against incorporating any supplementary physical exertion.
  Arms: Daily life
Behavioral: Functional general conditioning training — Training sessions were supervised by a certified instructor. Training was carried out at home with individually adjusted resistance depending on age and health. Participants typically performed 10-13 repetitions of a given exercise. 30-second rest intervals were used between exercises. As intended, the training was comprehensive, i.e. including muscles of the arms, legs, trunk, abdomen, chest, balance and flexibility exercises. Basic training equipment was used during the training.
  Arms: Functional general conditioning training

SUMMARY:
The aim of this clinical study is to examine the impact of physical activity on the physical and mental health of postmenopausal women, with a particular focus on the development of disability. The main questions this study aims to answer are:

1. Can physical activity programs (Nordic walking, Bungy Pump, strength training, functional general conditioning training) prevent loss of mobility, bone density and urinary incontinence, reduce the risk of falls, lower metabolic syndrome parameters, and improve cardiovascular endurance in postmenopausal women?
2. Do regular exercises improve cognitive functions, motivation, memory, visual coordination, mood, and quality of life in postmenopausal women?

Researchers will compare the test groups (Nordic Walking, Bungy Pump, strength training, functional general conditioning training) with the control group to determine whether physical activity brings benefits in terms of physical and mental health compared to no intervention.

Participants will:

Take part in a three-month physical activity program that includes Nordic walking, Bungy Pump exercises, functional general conditioning training and strength training, depending on the group.

The control group will not participate in any additional physical exercise program and will continue with their usual daily activities.

DETAILED DESCRIPTION:
This study will involve two testing phases (pre- and post-training). Prior to the first test, participants' physical activity will be measured over a period of seven days using POLAR accelerometers to evaluate the relationship between their daily physical activity and health. Each testing phase will last two days; on the first day, blood samples will be collected, and preliminary analyses of body composition and dietary records will be conducted. On the second day, physical fitness tests and psychological test swill be performed at the AWFiS Sports Exercise Laboratory in Gdańsk. Biological materials (serum) will be frozen and subsequently tested by contractors at the AWFiS Sports Genetics Laboratory. Participants will be required to maintain a dietary diary to record their dietary intake for the three days preceding the tests.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women over 60 years old (i.e. more than 12 months since their last menstrual cycle).

There were no contraindications to exercise after case reports and initial diagnosis.

Informed consent must be signed, agreeing to participate in research and physical exercise programs.

Exclusion Criteria:

* Uncontrolled high blood pressure. Rheumatoid arthritis. Type 2 diabetes. Are taking or have used antibiotics and/or antifungal therapy in the past 4 weeks.

Unwillingness to stick to a prescribed schedule.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2025-10-05 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Risk of Falls | From enrollment to the end of treatment at 3 months
  The Biodex Balance System (BBS) was used to assess the risk of fall test (RFT). The participants were asked to step on a platform in a bipedal stance with bare feet and open eyes looking forward to the BSS monitor to control the cursor, while their hands hung by their sides (hand support was not permitted). They were asked to stand straight, not to change their feet position, and only sway their body when necessary.
  Risk of Fall Test (RFT): The assessment of the dynamic bilateral stance was conducted on an unstable platform, where levels 6 to 2 were used. The test consisted of three measurements at intervals of 20 s of testing, and a break of 10 s. Prior to testing, the test procedure was explained. In this test, only the OSI was performed. This index was calculated through the degree of oscillation of the platform, where lower scores suggested better stability of th
Bone Density | From enrollment to the end of treatment at 3 months
  The densitometry test was conducted to assess the bone mineral density in women. The DEXA (dual-energy X-ray absorptiometry) technique was used, which allows precise measurements of bone mineral density. The measurement covered two key areas: the lumbar spine (L1-L4) and the femoral neck. The test involved positioning the patient on the densitometry table, where directed X-ray radiation passed through the tissues, enabling the calculation of bone mineral density in the designated areas. The entire process was painless and non-invasive, usually taking around 15-20 minutes. The participants were informed about the purpose of the test and that no special preparation was required. The results allowed for determining the bone mineral density in the selected areas, which served as the basis for assessing the risk of osteoporosis and other bone metabolic disorders.
Triglycerides (Metabolic syndrome Indicators) | From enrollment to the end of treatment at 3 months
  The level of triglycerides is one of the important indicators of human health. High or low levels of triglycerides in the blood can indicate certain health problems. The unit of TG is: mg/dl. Fasting venous blood samples will be collected after at least 12 hours of overnight stay. Blood will be collected in a Sarstedt S-Monovette tube without anticoagulants, but with the addition of coagulation factors to obtain serum. Serum samples will be processed according to standard laboratory procedures, aliquoted and stored at -80°C until analysis. Blood tests will be carried out by an external company.
Total cholesterol (Metabolic syndrome Indicators) | From enrollment to the end of treatment at 3 months
  Total cholesterol refers to the sum of cholesterol contained in all lipoproteins in the blood, and its serum concentration can be used as an indicator of lipid metabolism. The unit of TG is: mg/dl. Fasting venous blood samples will be collected after at least 12 hours of overnight stay. Blood will be collected in a Sarstedt S-Monovette tube without anticoagulants, but with the addition of coagulation factors to obtain serum. Serum samples will be processed according to standard laboratory procedures, aliquoted and stored at -80°C until analysis. Blood tests will be carried out by an external company.
High Density Lipoprotein Cholesterol (HDL-C) | From enrollment to the end of treatment at 3 months
  High-density lipoprotein (HDL) is one of the serum proteins, which is a complex lipoprotein composed of lipids, proteins and their regulators. HDL-C is a clinical test that represents the level of HDL in the blood. The unit of HDL-C is: mg/dl. Fasting venous blood samples will be collected after at least 12 hours of overnight stay. Blood will be collected in a Sarstedt S-Monovette tube without anticoagulants, but with the addition of coagulation factors to obtain serum. Serum samples will be processed according to standard laboratory procedures, aliquoted and stored at -80°C until analysis. Blood tests will be carried out by an external company.
non-High Density Lipoprotein Cholesterol (no-HDL-C) | From enrollment to the end of treatment at 3 months
  Non-high-density lipoprotein cholesterol (non-HDL-C) is the sum of cholesterol contained in lipoproteins other than HDL. Non-HDL cholesterol is a strong predictor of cardiovascular risk and can predict the progression of atherosclerosis. The unit of no-HDL-C is: mg/dl. Fasting venous blood samples will be collected after at least 12 hours of overnight stay. Blood will be collected in a Sarstedt S-Monovette tube without anticoagulants, but with the addition of coagulation factors to obtain serum. Serum samples will be processed according to standard laboratory procedures, aliquoted and stored at -80°C until analysis. Blood tests will be carried out by an external company.
Low Density Lipoprotein Cholesterol (LDL-C) | From enrollment to the end of treatment at 3 months
  Low-density lipoprotein cholesterol (LDL-C) is the main lipoprotein in fasting plasma. The content of LDL-C is related to the incidence and degree of cardiovascular disease, and is considered to be the main causative factor of atherosclerosis. LDL-C is measured in mg/dl. Fasting venous blood samples will be collected after at least 12 hours of overnight stay. Blood will be collected in a Sarstedt S-Monovette tube without anticoagulants, but with the addition of coagulation factors to obtain serum. Serum samples will be processed according to standard laboratory procedures, aliquoted and stored at -80°C until analysis. Blood tests will be carried out by an external company.
Fasting blood glucose (FBG) | From enrollment to the end of treatment at 3 months
  Fasting blood glucose (FBG) refers to the blood glucose value detected by the plasma collected before breakfast after fasting overnight (at least 8~10 hours without eating any food, except drinking water), which can reflect the function of pancreatic B cells, generally indicate the secretion function of basal insulin, and is the most commonly used detection index for diabetes. The unit of FBG is: mg/dl. Fasting venous blood samples will be collected after at least 12 hours of overnight stay. Blood will be collected in a Sarstedt S-Monovette tube without anticoagulants, but with the addition of coagulation factors to obtain serum. Serum samples will be processed according to standard laboratory procedures, aliquoted and stored at -80°C until analysis. Blood tests will be carried out by an external company.
Gait Speed | From enrollment to the end of treatment at 2 weeks
  In order to harmonize the pace measurement method, the 2019 Asian Sarcopenia Working Group recommends the time it takes to walk 6 meters at a normal pace from moving as a measure of average pace. The test is carried out in an inspection room that is more than 8 meters long. Crutches that participants normally use can also be used. The start and end of the 6-meter distance are clearly marked. Subjects stand with their toes touching the starting line, and after being instructed to move forward at their usual speed, subjects start walking, inspectors start timing, and when subjects fully cross the 6-meter mark with one foot, inspectors stop timing. The test is performed twice, recording the shortest time (in seconds) required to complete each distance. The smaller the value, the faster the walking speed, the better the physical ability.
Skeletal muscle index | From enrollment to the end of treatment at 2 weeks
  SMI in InBody is calculated as follows: SMI= sum of segmental muscle mass (two arms and two legs) ÷ height 2
Cognitive Abilities Assessment | From enrollment to the end of treatment at 3 months
  The study was conducted in a controlled laboratory using the Vienna Test System (VTS) with the Kognitron (COG) test to assess cognitive abilities. The participant, seated at a computer, performed tasks measuring working memory, attention, problem-solving, and decision-making. Clear instructions and a brief training phase ensured understanding of the tasks. The system recorded performance metrics such as reaction time and accuracy, automatically processing data to ensure objectivity. Test duration varied from several minutes to an hour, with detailed reports generated upon completion, ensuring standardized and reliable assessment.
Quality of Life | From enrollment to the end of treatment at 3 months
  The study utilized the WHOQOL-BREF questionnaire, a 26-item tool developed by the World Health Organization to assess quality of life across four domains: physical health, psychological well-being, social relationships, and environment. Participants, informed of the study's voluntary and anonymous nature, responded to statements using a Likert scale (1-5). Completing the questionnaire took 10-15 minutes, with researchers available for clarifications. Responses were analyzed per WHO guidelines, converting scores to a 0-100 scale for domain comparison. The results offer a comprehensive quality-of-life assessment, widely applicable in healthcare, psychology, and social research.
VO2max | From enrollment to the end of treatment at 3 months
  The EKBLOM-BAK test is a submaximal cycle ergometry test to estimate VO2max. After calibrating the ergometer and ensuring pre-test conditions (e.g., avoiding heavy meals, alcohol, and intense activity), the participant pedals at 60 rpm for 4 minutes at a workload targeting a heart rate of 110-140 bpm. Heart rate is averaged at specific intervals. The workload is then increased, and perceived exertion (RPE) is assessed. Adjustments to resistance depend on RPE ratings, with the test stopping if RPE exceeds 17. VO2max is estimated using collected data via a formula or an online tool. Suitable for individuals aged 20-86, the test provides reliable VO2max estimates.
Gait | From enrollment to the end of treatment at 3 months
  Gait analysis was conducted using the Zebris FDM-T treadmill, equipped with 10,240 force sensors (0.85 x 0.85 cm) to record reactive forces in three directions at 120 Hz. The treadmill's adjustable speed (0.2-22 km/h) enabled analysis at various paces. Participants walked barefoot, starting at 0.5 km/h with 0.3 km/h increments every 15 seconds, until determining their comfortable walking speed, followed by a 1-minute test.Spatiotemporal variability was assessed using the coefficient of variation (CV) for step length and time, with higher CV values indicating greater variability.
Static Balance | From enrollment to the end of treatment at 3 months
  Center of pressure (CoP) trajectory analysis provided insights into stability and balance. Static balance assessment included CoP sway area, path length, sway rate, and pressure distribution between feet. Participants stood barefoot with specific posture and completed three 20-second trials, with 30-second breaks between each.
Pelvic Floor Muscle Function | From enrollment to the end of treatment at 3 months
  The study consisted of two stages: completing the Incontinence Impact Questionnaire (IIQ) and evaluating pelvic floor muscle function using surface electromyography (sEMG) with biofeedback. In the first stage, participants completed the IIQ to assess the subjective impact of urinary incontinence on daily life. The data collected helped evaluate discomfort and limitations caused by incontinence. In the second stage, pelvic floor muscle function was assessed using sEMG with a vaginal electrode, measuring muscle activity at rest and during controlled contractions. Biofeedback training allowed participants to observe muscle activity in real time, helping improve control over pelvic floor muscle function.
Daily steps | Physical activity levels were monitored for 7 days prior to the test
  Assess physical activity levels over 7 days using the POLAR accelerometer, record daily steps.

SECONDARY OUTCOMES:
PEAK AWY | From enrollment to the end of treatment at 2 weeks
  Peak knee extension muscle strength. Using Biodex System 4 Pro™ dynamometers (Biodex Medical Systems, Inc.) Data collection using Compaq Desk Pro personal computers and Biodex software, using the Biodex standard protocol. After a standardized warm-up, the subject is positioned in the equipment as required by the manufacturer's manual (sitting position, arms hanging down along the body, hands holding the outside handle, torso, buttocks and subject thighs secured by straps, knee flexion to 90°). The test uses the scheme reported by Symons et al., with some modifications. The isometric muscle strength test was performed using three maximum contractions, each lasting 5 seconds with an interval of 30 seconds. Adjust the seat position according to the length of each subject's legs. Data were analyzed using the results of the dominant lower limbs. The greater the value of this index, the stronger the isometric contraction force of the knee extensor muscle.
PEAK TWD | From enrollment to the end of treatment at 2 weeks
  Peak knee flexor strength. Using Biodex System 4 Pro™ dynamometers (Biodex Medical Systems, Inc.) Data collection using Compaq Desk Pro personal computers and Biodex software, using the Biodex standard protocol. After a standardized warm-up, the subject is positioned in the equipment as required by the manufacturer's manual (sitting position, arms hanging down along the body, hands holding the outside handle, torso, buttocks and subject thighs secured by straps, knee flexion to 90°). The test uses the scheme reported by Symons et al., with some modifications. The isometric muscle strength test was performed using three maximum contractions, each lasting 5 seconds with an interval of 30 seconds. Adjust the seat position according to the length of each subject's legs. Data were analyzed using the results of the dominant lower limbs. The higher the value of this index, the stronger the isometric contraction force of knee flexor muscle.
Tandem Balance | From enrollment to the end of treatment at 2 weeks
  Participants used the "toe" stick to the "heel" in a straight-line walking way, with the fastest speed to complete 2 and 5 meters. The smaller the value, the faster the walking speed, which may represent better balance ability.
Arm strength index | From enrollment to the end of treatment at 2 weeks
  The arm strength HS was measured by a dynamometer, and the weight BM was measured in KG using a weight scale. Arm strength index calculation formula: HS/BM. A higher value for this indicator may mean greater muscle strength.
Skeletal Lean Mass | From enrollment to the end of treatment at 2 weeks
  Using the Octupole Bioimpedance InBody 720 analyzer (Biospace, Seoul, Korea), participants wore light clothing and no shoes. The calculation method of SLM is different from that of SMM. The SLM in InBody report paper is the sum of protein, body water, and extracosseous inorganic salts. The ideal SLM for men is 80% of standard body weight and 72% of standard body weight for women. A 10% move up or down is considered normal.
Pain pressure threshold (PPT) | From enrollment to the end of treatment at 3 months
  Pain pressure threshold (PPT) was assessed using the Medoc AlgoMed Seaweed Meter (Israel). PPT is the minimum pressure at which pressure turns into pain. Measurements are taken in a seated position on the back of the hand (between the thumb and forefinger) and the lateral arm (2/3 of the length of the arm). Stimulation was applied at a rate of 30 kPa/sec. When the pain is felt (PPT) measurement ends.
Electromyography | From enrollment to the end of treatment at 3 months
  After evaluating basic physical characteristics, women performed maximal voluntary contractions (MVCs) for EMG normalization. MVC measurements were taken using the Biodex System 4 dynamometer (Biodex Medical Systems Inc., USA) according to the manufacturer's guidelines. Settings included: 90° flexion and abduction of the shoulder, 90° flexion of the elbow with 45° shoulder flexion, 90° flexion of the knee and hip, and a neutral wrist position with 90° elbow flexion. Skin was prepared for EMG recording following SENIAM guidelines. Electrodes were placed on the dominant side muscles. EMG signals were collected with the Noraxon TeleMyo DTS system. Raw data were processed, rectified, smoothed, and normalized to MVC peak values for each individual, with results averaged over 3 attempts.
Postural Stability Test (PST) | From enrollment to the end of treatment at 3 months
  Subjects were subjected to a postural stability test (PST) using the Biodex Balance System (BBS). PST assesses postural stability using three metrics: OSI, APSI, and MLSI, with three 10-second trials on a stable platform. Higher scores indicate greater postural instability. Participants stand on the podium with their eyes wide open and their hands at their sides.
Spatial memory assessment | From enrollment to the end of treatment at 3 months
  The CORSI test was conducted using the Vienna Test System (VTS) software to assess the spatial memory of women. On the screen, nine irregularly positioned blocks appear. A hand-shaped cursor points to the blocks, which briefly light up, creating a sequence. After the sequence is completed, the participant must tap the same blocks in the same order. The test starts with three-block sequences, and the length of the sequences gradually increases to eight blocks. The test ends after three failed attempts with the eight-block sequence or after 18 trials. The test result measures visual memory, and the difficulty of the sequences increases with each subsequent trial. The test was conducted in a quiet environment to ensure the participants' comfort and focus.
Global Physical Activity Questionnaire (GPAQ) | From enrollment to the end of treatment at 3 months
  GPAQ involves completing a questionnaire about daily activity in three areas: work, transportation, and leisure. Participants report time spent on activities like walking, running, cycling, or physically demanding work. Responses are used to classify activity level (low, moderate, high).
Fall-related concerns | From enrollment to the end of treatment at 3 months
  The assessment using the Polish version of the Short FES-I (PL) involves the participant completing 7 questions about concerns related to falls in daily activities. The questionnaire evaluates the subjective perception of fall risk in various situations, such as walking upstairs, shopping, or walking outside. Participants respond to the questions, rating how insecure they feel in each situation using a Likert scale from 1 (very secure) to 4 (very insecure). The responses are summed, which allows for determining the level of fall-related concerns. The questionnaire is quick to complete and provides information about the participant's subjective perception of fall risk.
Cognitive Ability | From enrollment to the end of treatment at 3 months
  The Trail Making Test (TMT) is a tool used to assess cognitive functions, measuring the speed of information processing and cognitive flexibility. The test consists of two parts:
  Part A: The participant connects numbers (1-25) in ascending order by drawing a line between them. The time to complete the task is measured.
  Part B: The participant alternates between connecting numbers and letters (1-A-2-B-3-C…13-L), which requires greater cognitive flexibility. The time to complete this part is also measured.
  The test is conducted in a quiet, controlled environment. The participant receives clear in-structions before starting each part. The time taken for each part is measured, and the results are interpreted based on the total time. A longer time in Part B may indicate difficulties with executive functions. The test is a simple tool for assessing cognitive abilities in older adults.
30-Second Chair Stand | From enrollment to the end of treatment at 3 months
  Physical Fitness Test (SFT) levels in older adults were assessed by the 30-second chair standing test. Measures lower body strength. The participant stands as many times as possible in 30 seconds. Fewer than 8 stands indicate a risk zone.
Circumferences | From enrollment to the end of treatment at 3 months
  These tests provide a comprehensive assessment of an older adult's physical fitness, with spe-cific "risk zones" indicating potential areas of concern for strength, endurance, flexibility, and balance. The results help identify the need for targeted interventions or exercise programs.
  Measurement of waist, hip, arm, and calf circumferences in older adults is conducted to assess body composition and monitor physical health.
  Waist circumference is measured at the level of the navel, ensuring the measuring tape is ho-rizontal and fits snugly without compressing the skin. Hip circumference is measured at the widest point of the hips, with the tape kept level and not too tight.
  Arm circumference is measured at the midpoint between the shoulder joint and elbow, while calf circumference is taken at the widest point of the calf, ensuring the tape is neither too loo-se nor too tight.
  Measurements should be taken standing and breathing normally, with two repetitions and an average.
Forward Lean Test | From enrollment to the end of treatment at 3 months
  This test evaluates the ability to maintain balance while leaning the torso forward.
  Methodology: The participant stands in an upright position, with one arm extended forward, leaning against a wall. They then slowly lean their torso forward, aiming to maintain balance without touching the wall or the ground. The test is repeated three times, and the result is ba-sed on the best time the participant is able to maintain balance.
  Interpretation of Results: A longer time maintaining balance indicates good postural control, while difficulties in maintaining the position may suggest balance issues.
Sedentary time | From enrollment to the end of treatment at 3 months
  Description: Assess physical activity levels over 7 days using the POLAR accelerometer, record daily lying time, sitting time and standing time.Time Frame: Physical activity levels were monitored for 7 days prior to the test
Adiponectin (ADPN) | From enrollment to the end of treatment at 3 months
  Adiponectin (ADPN) is an endogenous bioactive peptide or protein secreted by adipocytes. Adiponectin is an insulin-sensitizing hormone that improves insulin resistance and arteriosclerosis, predicts the development of type II diabetes and coronary heart disease, and has demonstrated anti-diabetic, anti-atherotic and anti-inflammatory potential in clinical trials；the unit of adiponectin is: mg/dl. Blood collection and Adiponectin protein assay will be performed by an external company.
Hand Strength (HS) | From enrollment to the end of treatment at 3 months
  Description: HS was measured to estimate muscle strength and was performed with a hand dynamometer (SAEHAN Digital Hand Dynamometer, SAEHAN, Changwon, Korea). During the HS test, participants had to hold the dynamometer in their hand with the arm stretched parallel to the body while being instructed to stand upright. This measure was performed three times on the dominant hand with a rest interval of 1 min between measurements; finally, the best performance was used as the maximum peak (PK) of HS (in kg). The statistical analysis also included mean peak (mean PK). The higher the grip strength value, the greater the muscle strength, the better the physical ability.
Skeletal Muscle Mass | From enrollment to the end of treatment at 3 months
  Description: Using the Octupole Bioimpedance InBody 720 analyzer (Biospace, Seoul, Korea), participants wore light clothing and no shoes. The higher the number, the more muscle the human body has. The ideal skeletal muscle content for men is 47% of standard body weight and 42% of standard body weight for women. A 10% move up or down is considered normal.
Myostatin | From enrollment to the end of treatment at 3 months
  Myostatin is a protein whose units are the same as those of other proteins, usually expressed in moles (mol/L). The MAGPIX platform enables multiplex tests, which allow for multi-parameter detection of several to several dozen analytes in a single sample of small volume (~40ul). The MAGPIX (xMAP®) system is based on the principles of the ELISA test and uses the technology of paramagnetic microspheres coated with antibodies. One panel- Page 5 of 9 [DRAFT] allows for simultaneous determination of several to several dozen markers in each sample. ELISA (enzyme-linked immunosorbent assay) is an immunoenzymatic test used to detect and quantify proteins contained in the tested sample, such as antibodies or protein antigens. The ELISA technique is widely used in biomedical research, both scientific and diagnostic. It is a fast, accurate and easy to perform method. Consumables: nitrile gloves, pipette tips 10-200ul, pipette tips 100-1000ul, eppendorff tubes, other (falcon tubes, etc.)
Irisin | From enrollment to the end of treatment at 3 months
  The unit of irisin is molecular weight and its value is 298.25. The MAGPIX platform enables multiplex tests, which allow for multi-parameter detection of several to several dozen analytes in a single sample of small volume (~40ul). The MAGPIX (xMAP®) system is based on the principles of the ELISA test and uses the technology of paramagnetic microspheres coated with antibodies. One panel allows for simultaneous determination of several to several dozen markers in each sample. ELISA (enzyme-linked immunosorbent assay) is an immunoenzymatic test used to detect and quantify proteins contained in the tested sample, such as antibodies or protein antigens. The ELISA technique is widely used in biomedical research, both scientific and diagnostic. It is a fast, accurate and easy to perform method. Consumables: nitrile gloves, pipette tips 10-200ul, pipette tips 100-1000ul, eppendorff tubes, other (falcon tubes, lignin, etc.).
BDNF | From enrollment to the end of treatment at 3 months
  BDNF (brain-derived neurotrophic factor) assay unit is mainly pg/mL. The MAGPIX platform enables multiplex tests, which allow for multi-parameter detection of several to several dozen analytes in a single sample of small volume (~40ul). The MAGPIX (xMAP®) system is based on the principles of the ELISA test and uses the technology of paramagnetic microspheres coated with antibodies. One panel allows for simultaneous determination of several to several dozen markers in each sample. ELISA (enzyme-linked immunosorbent assay) is an immunoenzymatic test used to detect and quantify proteins contained in the tested sample, such as antibodies or protein antigens. The ELISA technique is widely used in biomedical research, both scientific and diagnostic. It is a fast, accurate and easy to perform method. Consumables: nitrile gloves, pipette tips 10-200ul, pipette tips 100-1000ul, eppendorff tubes, other (falcon tubes, lignin, etc.).
Arm strength index II | From enrollment to the end of treatment at 2 weeks
  The arm flexor strength HS was measured by a dynamometer, and the BMI was measured in KG/m2. Arm strength index calculation formula: HS/BMI. A higher value for this indicator may mean greater muscle strength.
Knee extensor strength index | From enrollment to the end of treatment at 2 weeks
  The knee extensor strength HS was measured using a dynamometer, and the weight BM was measured in kg using a weight scale. Knee extensor strength index calculation formula: HS/BM. A higher value for this indicator may mean greater muscle strength.
Knee flexor strength index | From enrollment to the end of treatment at 2 weeks
  The knee flexor strength HS was measured using a dynamometer, and the weight BM was measured in kg using a weight scale. Knee flexor strength index calculation formula: HS/BM. A higher value for this indicator may mean greater muscle strength.
Pain tolerance (PTOL) | From enrollment to the end of treatment at 3 months
  Pain tolerance (PTOL) was assessed using the Medoc AlgoMed Seaweed Meter (Israel). PTOL is the maximum pain intensity a person can withstand. Measurements are taken in a seated position on the back of the hand (between the thumb and forefinger) and the lateral arm (2/3 of the length of the arm). Stimulation was applied at a rate of 30 kPa/sec. Measurement ends when the participant can no longer tolerate stimulation.
Pain intensity score | From enrollment to the end of treatment at 3 months
  Participants rated pain intensity using the VAS scale (0-10). The higher the score, the greater the level of pain.
Limits of Stability Test (LOS) | From enrollment to the end of treatment at 3 months
  Subjects were subjected to a limits of stability Test (LOS) using the Biodex Equilibrium System (BBS). In the LOS test, the platform is stable and participants transfer their body weight to move the cursor from the central target to the peripheral target. This test measures the maximum angle that the body can reach vertically without losing its balance. Three trials were conducted.
International Physical Activity Questionnaire (IPAQ) | From enrollment to the end of treatment at 3 months
  IPAQ evaluates activity over the past 7 days, focusing on vigorous and moderate activity and sitting time. Based on responses, total activity time is calculated and classified (low, moderate, high).
Arm Curl | From enrollment to the end of treatment at 3 months
  Physical Fitness Test (SFT) levels in older adults were assessed by arm curl test. Measures upper body strength. The participant performs as many curls as possible in 30 seconds with a weight. Fewer than 11 curls indicate a risk zone.
6-Minute Walk | From enrollment to the end of treatment at 3 months
  Physical Fitness Test (SFT) levels in older adults were assessed by 6-minute walk. Measures aerobic endurance. The participant walks as far as possible in 6 minutes. Walking less than 350 yards indicates a risk zone.
Chair Sit-and-Reach | From enrollment to the end of treatment at 3 months
  Physical Fitness Test (SFT) levels in older adults were assessed by chair sit-and-reach. Measures lower body flexibility. A negative distance of more than 4 inches for men or 2 inches for women indicates a risk zone.
Back Scratch | From enrollment to the end of treatment at 3 months
  Physical Fitness Test (SFT) levels in older adults were assessed by back scratch. Measures upper body flexibility. A gap of more than 4 inches for men or 2 inches for women indicates a risk zone.
8-Foot Up-and-Go | From enrollment to the end of treatment at 3 months
  Physical Fitness Test (SFT) levels in older adults were assessed by 8-Foot Up-and-Go. Measures agility. A time over 9 seconds indicates a risk zone.
Leptin | From enrollment to the end of treatment at 3 months
  Leptin is a hormone secreted by adipose tissue, and its amount in serum is proportional to the size of the animal's adipose tissue. The negative feedback mechanism of leptin in serum can regulate the energy balance of organisms as well as body weight. Leptin is measured in pg/ml. The level of leptin will be determined using the MAGPIX fluorescence detection system (Luminex Corp., Austin, TX, USA) and the Luminex human magnetic assay 6-Plex according to the manufacturer's protocol. Data acquisition and analysis will be performed using xPONENT software and Quantist Luminex from Bio-Techne (Luminex Corp., Austin, TX, USA). Blood tests will be carried out by an external company.
Resistin | From enrollment to the end of treatment at 3 months
  Resistin is a cysteine-rich fat-derived peptide hormone that functions as a pro-inflammatory cytokine and can act as an important node in inflammatory diseases. Leptin is measured in pg/ml. The level of leptin will be determined using the MAGPIX fluorescence detection system (Luminex Corp., Austin, TX, USA) and the Luminex human magnetic assay 6-Plex according to the manufacturer's protocol. Data acquisition and analysis will be performed using xPONENT software and Quantist Luminex from Bio-Techne (Luminex Corp., Austin, TX, USA).

OTHER OUTCOMES:
Body Fat Mass | From enrollment to the end of treatment at 2 weeks
  Using the Octupole Bioimpedance InBody 720 analyzer (Biospace, Seoul, Korea), participants wore light clothing and no shoes.The higher the value of this index, the higher the body fat content.
Fat-Free Mass | From enrollment to the end of treatment at 2 weeks
  Using the Octupole Bioimpedance InBody 720 analyzer (Biospace, Seoul, Korea), participants wore light clothing and no shoes. The higher the value of this index, the heavier the body weight without fat.
BMI | From enrollment to the end of treatment at 2 weeks
  Using the Octupole Bioimpedance InBody 720 analyzer (Biospace, Seoul, Korea), participants wore light clothing and no shoes. The average person's BMI is usually between 18 and 23.
Bifidobacterium | From enrollment to the end of treatment at 3 months
  Bifidobacteria are beneficial bacteria in the gut, and testing can determine their relative numbers in the gut flora. Microbiome testing will be performed at the AWFiS Sports Genetics Laboratory. DNA was isolated using a Bead Ruptor 24 Elite homogenizer and a QIAamp PowerFecal Pro DNA Kit (Qiagen) according to the manufacturer's procedure. The quality and quantity of the separated material will be checked on a NanoDrop 1000 spectrophotometer (Thermo Scientific), Qubit 4.0 fluorometer (ThermoFisher). Sequencing in PE mode (2x150 bp) will be performed on the NovaSeq platform (Illumina).
The vitamin D3 level test | From enrollment to the end of treatment at 3 months
  The blood vitamin D3 level test in women was conducted to assess its concentration in the body. Blood samples for analysis were taken from the antecubital vein using standard sample collection procedures. The sample was then sent to the laboratory, where the level of 25-hydroxyvitamin D (25(OH)D) was measured, as it is the primary indicator for evaluating vitamin D status in the body. The tests were performed using an immunoenzymatic method, ensuring precise and reliable results.
Blood sodium content test | From enrollment to the end of treatment at 3 months
  The amount of sodium in the blood is measured using the potentiometric method. The unit of detection is pg/mL. Blood is drawn in a fasting state, and sodium levels in the blood are measured using the potentiometric method of selective electrodes. Results are automatically recorded and evaluated according to clinical norms. Blood tests will be carried out by an external company.
IL-6 | From enrollment to the end of treatment at 3 months
  The unit of IL-6 (interleukin-6) is (pg/mL). Fasting venous blood samples will be collected after a minimum of 12 hours overnight. Blood will be collected in Sarstedt S-Monovette tubes without anticoagulants but with the addition of coagulation factors to obtain serum. Serum samples will be processed according to standard laboratory procedures, aliquoted and stored at -80°C until analysis. Levels of inflammatory markers CRP, IL-6 and TNF-alpha will be determined using the MAGPIX fluorescence detection system (Luminex Corp., Austin, TX, USA) and the Luminex Human Magnetic Assay 6-Plex according to the manufacturer's protocols. Data acquisition and analysis will be performed using xPONENT software and Quantist Luminex by Bio-Techne (Luminex Corp., Austin, TX, USA).
CRP | From enrollment to the end of treatment at 3 months
  CRP is an acute phase reaction protein, the unit of CRP is: mg/L. Blood collection and C-reactive protein assay will be performed by an external company
TNF-α | From enrollment to the end of treatment at 3 months
  TNF-α (tumor necrosis factor-α) has two molecular weights: 17kD monomer form and 51kD trimer form . According to the molecular weight, the concentration unit of TNF-α can be converted. For example, in the monomer form of TNF-α, 1ug is approximately equal to 0.06nmol; In trimer form TNF-α, 1ug is equal to approximately 0.02nmol.
  Serum samples will be processed according to standard laboratory procedures, aliquoted and stored at -80°C until analysis. Levels of inflammatory markers CRP, IL-6 and TNF-alpha will be determined using the MAGPIX fluorescence detection system (Luminex Corp., Austin, TX, USA) and the Luminex Human Magnetic Assay 6-Plex according to the manufacturer's protocols. Data acquisition and analysis will be performed using xPONENT software and Quantist Luminex by Bio-Techne (Luminex Corp., Austin, TX, USA).
Assessment of food types and quantities | From enrollment to the end of treatment at 3 months
  The type and number of things were assessed based on the dietary diaries kept by the study participants using dietary analysis software. The nutritional analysis in the Nuvero program is based on entering data from a diet diary and assessing the type and amount of food ingested based on the nutritional needs of the person being examined. The process begins with the collection of detailed information about the products and dishes consumed, which are recorded in a dietary diary kept by the person being examined. This information should include: the type and quantity of food consumed. The collected data is entered into the Nuvero program, which selects the products and dishes that most closely match the entries in the journal from the available database. If necessary, modifications to the composition of the dish or the method of preparation should be considered to ensure the accuracy of the analysis.
Visuomotor coordination (average deviation from the correct angle) | From enrollment to the end of treatment at 3 months
  The visuomotor coordination test, conducted using the SMK test in the Vienna Test System (VTS), assesses the ability to control spatial objects. A 3D room appears on the screen with a green "T" and a yellow circular segment. The segment moves in three ways: tilting, horizontal motion, and front-to-back, while changing size. The participant must use joysticks or foot pedals to control the segment so it stands upright, touching the green "T" intersection, and matches the size of the vertical bar. The correct metric for testing is the average deviation of the moving mark from the correct angle. Additionally, consistency is assessed by calculating the distribution of deviations over time.
Spinal Pain Assessment (Neck Disability Index) | From enrollment to the end of treatment at 3 months
  The impact of spinal cord pain on daily functioning was assessed by the Neck Disability Index (NDI). Participants were instructed to complete questionnaires assessing pain and its impact on physical, emotional, and social functioning. The NDI contains 10 questions on daily activities, with scores ranging from 0 (no problem) to 5 (severely limited). After completing the questionnaire, the results are converted to a percentage score to determine the degree of disability. Assessment is useful in diagnosing and monitoring treatment progress.
Reaction speed assessment | From enrollment to the end of treatment at 3 months
  Reaction speed assessment using the Blink system. Participants stand in front of a Blink device with lights around the wheels. The goal is to press the corresponding button to extinguish the lit light as soon as possible. The test lasts 1 minute, during which the indicator lights up randomly. Participants turn off the lights by pressing the correct buttons, and the reaction time is from the time the lights are on to off. The system automatically records the reaction time taken by the participant to turn off the light each time and the number of times the light is on. The speed of the participant's reaction was assessed by calculating the sum of the reaction time and the total number of light ons.
Range of motion | From enrollment to the end of treatment at 3 months
  Range of motion was measured for shoulder and hip joints using a long-arm goniometer. For the shoulder, the participant sat with arms relaxed, and the goniometer was placed on the shoulder joint. Flexion and extension of the arm were performed, aiming for full motion. The measurement was repeated three times for accuracy. For the hip, the participant lay on their side with the knee slightly bent. The goniometer was placed on the hip joint while flexion and extension of the leg were performed. This measurement was also repeated three times. Each test was performed with attention to joint stability and proper goniometer positioning.
Skinfold thickness measurement | From enrollment to the end of treatment at 3 months
  The skinfold thickness measurement in women was conducted to assess the subcutaneous tissue thickness at selected body sites: the triceps, biceps, subscapular region, torso, abdomen, thigh, and calf. The measurement was performed using a skinfold caliper, following standardized procedures to ensure accuracy and repeatability of the results. The skinfold was pinched using the thumb and index finger at the designated site, separating the skin and subcutaneous tissue from the underlying muscles. The caliper was applied perpendicular to the fold approximately 1 cm from the pinch site. The measurement was read after a few seconds to allow for a stable reading. Each measurement was repeated three times at each site, and the mean value of these measurements was used for analysis. The assessment was conducted under consistent environmental conditions, with participants maintaining a standardized body position to minimize external factors influencing the results.
Mood | From enrollment to the end of treatment at 3 months
  Women's emotions were studied using the UMACL (UWIST Emotional Adjective List) questionnaire to assess their emotions in three dimensions: emotional tension, energy, and pleasure. The questionnaire consists of a set of adjectives, and participants rate them on a four-point scale based on how they are currently feeling, ranging from "absolutely not" to "definitely yes." Participants were informed of the purpose of the study and were asked to complete the questionnaire in a calm environment, remaining anonymous to ensure free and honest responses. The completion time is about 5-10 minutes. The results are analysed to obtain numerical values for each of the three dimensions, thus being able to assess their mood at that time. The scale is usually scored on a scale from 0 to 5, with higher scores indicating a better emotional state in the dimensions of positive emotions (e.g., "happy", "excited", etc.), and higher scores in the dimensions of negative emotions (e.g., "frustration", "anxiety
Assessment of exercise motivation | From enrollment to the end of treatment at 3 months
  The study of women using the EFST Physical Activity Motivation Questionnaire (MPAM-r) aimed to evaluate motivation for physical activity in various contexts. The MPAM-r consists of questions measuring different aspects of motivation, such as intrinsic motivation (e.g., improving fitness, health), extrinsic motivation (e.g., improving appearance), and amotivation. Participants were asked to rate statements regarding their motivation for physical activity on a scale from 1 (strongly disagree) to 5 (strongly agree). The questionnaire was completed individually in a quiet, comfortable environment, with participants informed about the study's purpose and the assurance of anonymity to encourage honest responses. Completing the questionnaire took approximately 10-15 minutes. The results allowed for the evaluation of women's motivation for physical activity and the identification of factors influencing their decisions.
Assessment of self-esteem level | From enrollment to the end of treatment at 3 months
  The study of women using the Rosenberg Self-Esteem Scale (SES) aimed to assess their self-esteem level. The questionnaire consists of 10 statements to which participants respond, evaluating them on a four-point Likert scale, from "strongly disagree" to "strongly agree." The scale includes questions regarding perceived self-worth, self-confidence, and general attitude toward oneself. The study was conducted in comfortable conditions, in a quiet and private setting, to ensure participants' comfort and the ability to provide honest responses. Participants were informed about the purpose of the study, and anonymity was guaranteed to ensure reliable and accurate results. The time to complete the questionnaire was approximately 5-10 minutes. The results allowed for the assessment of women's self-esteem level. The scale is scored on 4 levels, with a minimum score of 1 point and a maximum score of 4 points, and the total score ranges from 10-40 points, with higher scores and higher self-estee
Lactobacillus | From enrollment to the end of treatment at 3 months
  Lactobacilli and others are beneficial bacteria in the gut, and testing can determine their relative numbers in the gut flora. Microbiome testing will be performed at the AWFiS Sports Genetics Laboratory. DNA was isolated using a Bead Ruptor 24 Elite homogenizer and a QIAamp PowerFecal Pro DNA Kit (Qiagen) according to the manufacturer's procedure. The quality and quantity of the separated material will be checked on a NanoDrop 1000 spectrophotometer (Thermo Scientific), Qubit 4.0 fluorometer (ThermoFisher). Sequencing in PE mode (2x150 bp) will be performed on the NovaSeq platform (Illumina).
Test of potassium content in the blood | From enrollment to the end of treatment at 3 months
  The amount of potassium in the blood is measured using the potentiometric method. The unit of detection is pg/mL. Blood is drawn on an empty stomach and potassium levels in the blood are measured using the potentiometric method of selective electrodes. Results are automatically recorded and evaluated according to clinical norms. Blood tests will be carried out by an external company.
Creatinine | From enrollment to the end of treatment at 3 months
  The study used an automated hematology analyzer to analyze blood morphology. Blood is drawn on a fasting state, and the amount of creatinine in the blood is measured using spectrophotometry to assess the absorption of light at a specific wavelength. The unit of detection is umol/L. Blood tests will be carried out by an external company.
Creatine kinase | From enrollment to the end of treatment at 3 months
  The study used an automated hematology analyzer to analyze blood morphology. Blood is drawn on a fasting state, and creatine kinase levels in the blood are measured using spectrophotometric assessment of light absorption at specific wavelengths. The unit of detection is umol/L. Blood tests will be carried out by an external company.
Uric acid | From enrollment to the end of treatment at 3 months
  The study used an automated hematology analyzer to analyze blood morphology. Blood is drawn on an empty stomach and the amount of uric acid in the blood is measured using spectrophotometry to assess light absorption at specific wavelengths. The unit of detection is umol/L. Blood tests will be carried out by an external company.
Albumin | From enrollment to the end of treatment at 3 months
  The study used an automated hematology analyzer to analyze blood morphology. Blood is drawn on an empty stomach and the amount of uric acid in the blood is measured using spectrophotometry to assess light absorption at specific wavelengths. The unit of detection is umol/L. Blood tests will be carried out by an external company.
Total protein | From enrollment to the end of treatment at 3 months
  The study used an automated hematology analyzer to analyze blood morphology. Blood is drawn on an empty stomach and the total protein content in the blood is measured using spectrophotometry to assess light absorption at specific wavelengths. The unit of detection is umol/L. Blood tests will be carried out by an external company.
ALT | From enrollment to the end of treatment at 3 months
  The study used an automated hematology analyzer to analyze blood morphology. Blood is drawn on an empty stomach and ALT levels in the blood are measured using spectrophotometry to assess light absorption at specific wavelengths. The unit of detection is umol/L. Blood tests will be carried out by an external company.
AST | From enrollment to the end of treatment at 3 months
  The study used an automated hematology analyzer to analyze blood morphology. Blood is drawn on an empty stomach and AST levels in the blood are measured using spectrophotometry to assess light absorption at specific wavelengths. The unit of detection is umol/L. Blood tests will be carried out by an external company.
Test of calcium content in the blood | From enrollment to the end of treatment at 3 months
  The study used an automated hematology analyzer to analyze blood morphology. Blood is drawn on an empty stomach and the amount of calcium in the blood is measured using spectrophotometry to assess the absorption of light at a specific wavelength. The unit of detection is umol/L. Blood tests will be carried out by an external company.
Magnesium content test in the blood | From enrollment to the end of treatment at 3 months
  The study used an automated hematology analyzer to analyze blood morphology. Blood is drawn on an empty stomach and the amount of magnesium in the blood is measured using spectrophotometry to assess the absorption of light at a specific wavelength. The unit of detection is umol/L. Blood tests will be carried out by an external company.
Red blood cells | From enrollment to the end of treatment at 3 months
  The study includes blood morphology tests. Blood is drawn on a fasting state and the number of red blood cells is analyzed using an automated hematology analyzer. Results are automatically recorded and evaluated according to clinical norms. Blood tests will be carried out by an external company.
Leukocytes | From enrollment to the end of treatment at 3 months
  The study includes blood morphology tests. Blood is drawn on an empty stomach and the number of white blood cells is analyzed using an automated hematology analyzer. Results are automatically recorded and evaluated according to clinical norms. Blood tests will be carried out by an external company.
Platelets | From enrollment to the end of treatment at 3 months
  The study includes blood morphology tests. Blood is drawn on an empty stomach and the number of platelets is analyzed using an automated hematology analyzer. Results are automatically recorded and evaluated according to clinical norms. Blood tests will be carried out by an external company.
Hemoglobin level | From enrollment to the end of treatment at 3 months
  The study includes blood morphology tests. Blood is drawn on a fasting state, and the amount of hemoglobin levels is analyzed using an automated hematology analyzer. Results are automatically recorded and evaluated according to clinical norms. Blood tests will be carried out by an external company.
Food calorie assessment | From enrollment to the end of treatment at 3 months
  Caloric content assessment based on dietary diaries kept by study participants using dietary analysis software. The nutritional analysis in the Nuvero program is based on data input from a dietary diary and an assessment of the caloric content of the ingested food based on the nutritional needs of the person being examined. The process begins with the collection of detailed information about the products and dishes consumed, which are recorded in a dietary diary kept by the person being examined. Depending on the type of food ingested, the portion size, the calories of the food are calculated through the Nuvero program.
Visuomotor coordination (deviations from horizontal/vertical lines) | From enrollment to the end of treatment at 3 months
  The visuomotor coordination test, conducted using the SMK test in the Vienna Test System (VTS), assesses the ability to control spatial objects. A 3D room appears on the screen with a green "T" and a yellow circular segment. The segment moves in three ways: tilting, horizontal motion, and front-to-back, while changing size. The participant must use joysticks or foot pedals to control the segment so it stands upright, touching the green "T" intersection, and matches the size of the vertical bar. The correct metric for testing is the deviations from horizontal/vertical lines. Additionally, consistency is assessed by calculating the distribution of deviations over time.
Visuomotor coordination (time spent in the ideal range) | From enrollment to the end of treatment at 3 months
  The visuomotor coordination test, conducted using the SMK test in the Vienna Test System (VTS), assesses the ability to control spatial objects. A 3D room appears on the screen with a green "T" and a yellow circular segment. The segment moves in three ways: tilting, horizontal motion, and front-to-back, while changing size. The participant must use joysticks or foot pedals to control the segment so it stands upright, touching the green "T" intersection, and matches the size of the vertical bar. The correct metric for testing is the time spent in the ideal range. Additionally, consistency is assessed by calculating the distribution of deviations over time.
Spinal Pain Assessment (Oswestry Disability Index) | From enrollment to the end of treatment at 3 months
  The impact of spinal cord pain on daily functioning was assessed by the Oswestry Disability Index. Participants were instructed to complete questionnaires assessing pain and its impact on physical, emotional, and social functioning. The Oswestry index has 10 sections on pain, mobility, work, and daily activities and is rated from 0 to 5. After completing both questionnaires, the results were converted to a percentage score to determine the degree of disability. Assessment is useful in diagnosing and monitoring treatment progress.
Faecalibacterium | From enrollment to the end of treatment at 3 months
  Description: Faecalibacterium is a genus of bacteria that is one of the most important components of a healthy human gut microbiota. Microbiome testing will be performed at the AWFiS Sports Genetics Laboratory. DNA was isolated using a Bead Ruptor 24 Elite homogenizer and a QIAamp PowerFecal Pro DNA Kit (Qiagen) according to the manufacturer's procedure. The quality and quantity of the separated material will be checked on a NanoDrop 1000 spectrophotometer (Thermo Scientific), Qubit 4.0 fluorometer (ThermoFisher). Sequencing in PE mode (2x150 bp) will be performed on the NovaSeq platform (Illumina).
Enterobacteriaceae | From enrollment to the end of treatment at 3 months
  Enterobacteriaceae is a family of Gram-negative bacteria that are commonly found in the environment, as well as in the human gastrointestinal tract. Microbiome testing will be performed at the AWFiS Sports Genetics Laboratory. DNA was isolated using a Bead Ruptor 24 Elite homogenizer and a QIAamp PowerFecal Pro DNA Kit (Qiagen) according to the manufacturer's procedure. The quality and quantity of the separated material will be checked on a NanoDrop 1000 spectrophotometer (Thermo Scientific), Qubit 4.0 fluorometer (ThermoFisher). Sequencing in PE mode (2x150 bp) will be performed on the NovaSeq platform (Illumina).
Sleep Quality | From enrollment to the end of treatment at 3 months
  The Pittsburgh Sleep Quality Index (PSQI) is a tool used to assess sleep quality over the past month based on 19 self-reported questions. It analyzes seven components: subjective sleep quality, latency, duration, efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each component is rated on a scale of 0-3, and the total score (0-21) determines sleep quality - a score ≤5 indicates good sleep quality, while a score >5 suggests sleep problems. PSQI is widely used in scientific and clinical research, particularly in the diagnosis of insomnia and mental health disorders, and is recognized as a reliable and repeatable tool.

CONTACTS AND LOCATIONS:
Overall Officials: Zbigniew Ossowski, PHD, Study Chair — AKADEMIA WYCHOWANIA FIZYCZNEGO I SPORTU; Yangjun Liu, PHD, Principal Investigator — Chengdu University of Traditional Chinese Medicine
Locations (1):
- Gdansk University of Physical Education and Sport, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
There are some privacy concerns.

REFERENCES:
- [Background] Ricci NA, Cunha AIL. Physical Exercise for Frailty and Cardiovascular Diseases. Adv Exp Med Biol. 2020;1216:115-129. doi: 10.1007/978-3-030-33330-0_12. PMID 31894552
- [Background] Gallardo-Gomez D, Del Pozo-Cruz J, Noetel M, Alvarez-Barbosa F, Alfonso-Rosa RM, Del Pozo Cruz B. Optimal dose and type of exercise to improve cognitive function in older adults: A systematic review and bayesian model-based network meta-analysis of RCTs. Ageing Res Rev. 2022 Apr;76:101591. doi: 10.1016/j.arr.2022.101591. Epub 2022 Feb 17. PMID 35182742
- [Background] Todhunter-Brown A, Hazelton C, Campbell P, Elders A, Hagen S, McClurg D. Conservative interventions for treating urinary incontinence in women: an Overview of Cochrane systematic reviews. Cochrane Database Syst Rev. 2022 Sep 2;9(9):CD012337. doi: 10.1002/14651858.CD012337.pub2. PMID 36053030
- [Background] Hopewell S, Adedire O, Copsey BJ, Boniface GJ, Sherrington C, Clemson L, Close JC, Lamb SE. Multifactorial and multiple component interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2018 Jul 23;7(7):CD012221. doi: 10.1002/14651858.CD012221.pub2. PMID 30035305
- [Background] Huynh E, Wiley E, Noguchi KS, Fang H, Beauchamp MK, MacDonald MJ, Tang A. The effects of aerobic exercise on cardiometabolic health in postmenopausal females: A systematic review and meta-analysis of randomized controlled trials. Womens Health (Lond). 2024 Jan-Dec;20:17455057241290889. doi: 10.1177/17455057241290889. PMID 39431435
- [Background] Neilson HK, Conroy SM, Friedenreich CM. The Influence of Energetic Factors on Biomarkers of Postmenopausal Breast Cancer Risk. Curr Nutr Rep. 2013 Dec 15;3(1):22-34. doi: 10.1007/s13668-013-0069-8. eCollection 2014. PMID 24563822
- [Background] Remie CME, Janssens GE, Bilet L, van Weeghel M, Duvivier BMFM, de Wit VHW, Connell NJ, Jorgensen JA, Schomakers BV, Schrauwen-Hinderling VB, Hoeks J, Hesselink MKC, Phielix E, Houtkooper RH, Schrauwen P. Sitting less elicits metabolic responses similar to exercise and enhances insulin sensitivity in postmenopausal women. Diabetologia. 2021 Dec;64(12):2817-2828. doi: 10.1007/s00125-021-05558-5. Epub 2021 Sep 12. PMID 34510226
- [Background] Ra JS, Kim H. Combined Effects of Unhealthy Lifestyle Behaviors on Metabolic Syndrome among Postmenopausal Women. Healthcare (Basel). 2021 Jul 5;9(7):848. doi: 10.3390/healthcare9070848. PMID 34356226
- [Background] Teraz K, Kalc M, Peskar M, Pisot S, Simunic B, Pisot R, Pori P. Sarcopenia, obesity, and their association with selected behavioral factors in active older adults. Front Physiol. 2023 Feb 23;14:1129034. doi: 10.3389/fphys.2023.1129034. eCollection 2023. PMID 36909226
- [Background] Partridge L, Deelen J, Slagboom PE. Facing up to the global challenges of ageing. Nature. 2018 Sep;561(7721):45-56. doi: 10.1038/s41586-018-0457-8. Epub 2018 Sep 5. PMID 30185958
- [Background] Ossowski ZM, Skrobot W, Aschenbrenner P, Cesnaitiene VJ, Smaruj M. Effects of short-term Nordic walking training on sarcopenia-related parameters in women with low bone mass: a preliminary study. Clin Interv Aging. 2016 Nov 30;11:1763-1771. doi: 10.2147/CIA.S118995. eCollection 2016. PMID 27942207